CLINICAL TRIAL: NCT06778291
Title: Patients Comfort During Highflow Oxygen Therapy With Asymmetrical Prongs
Acronym: COMFOXY-1
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Annalisa Boscolo, Professor, University of Padova
Other Study IDs: COMFOXY-1
Record Dates: First submitted 2025-01-07; First posted 2025-01-16 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Failure
Keywords: high flow oxygen therapy; oxygen therapy
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OCCLUDING HFNC then SMALLER HFNC: Randomization will be performed immediately after the enrollment of the patient, before starting HFNC support. All patients will receive HFNC therapy through the asymmetrical interface Optiflow® Duet system (Fisher & Paykel Healthcare, Auckland, New Zealand). According to a software-generated blocked random sequence, patients will be assigned to the larger cannula treatment and then the smaller cannula treatment or viceversa.
- SMALLER HFNC then OCCLUDING HFNC: Randomization will be performed immediately after the enrollment of the patient, before starting HFNC support. All patients will receive HFNC therapy through the asymmetrical interface Optiflow® Duet system (Fisher & Paykel Healthcare, Auckland, New Zealand). According to a software-generated blocked random sequence, patients will be assigned to the larger cannula treatment and then the smaller cannula treatment or viceversa.

SUMMARY:
High-flow nasal cannula (HFNC) is a respiratory support device widely used to manage acute respiratory failure (ARF) and recommended in different patient populations according to the last European Respiratory Society and European Society of Intensive Care Medicine guidelines. HFNC delivers heated and humidified oxygen that facilitates airway secretion clearance, and its use is associated with improvement of oxygenation and reduction of airway dead space compared to standard oxygen therapy. Finally, all these beneficial effects result in a greater comfort experienced by the patient, as compared either to standard oxygen therapy or non-invasive ventilation.

DETAILED DESCRIPTION:
Recently, a new HFNC interface using asymmetrical prongs (Optiflow® Duet system, Fisher & Paykel Healthcare, Auckland, New Zealand) was approved for clinical practice. Unlike nasal cannulas with equally sized prongs, asymmetrical prongs deliver different flow rates between the two nostrils. Bench studies have demonstrated that the asymmetrical configuration resulted in higher positive end-expiratory pressure (PEEP) and accelerated clearance of the anatomical dead space.

In a recent physiological cross-over study, randomizing 20 intensive care unit (ICU) patients with post-extubation hypoxemic ARF to the asymmetrical or symmetrical interface, the use of asymmetrical HFNCs, despite showing similar performances in terms of lung aeration, ventilatory efficiency, gas exchange, and inspiratory effort, was associated with improved patient comfort, compared to standard HFNC interface. However, the study population included mostly patients with moderate hypoxemic ARF and near-normal respiratory rate, while only few patients suffered severe hypoxemia or tachypnea.

Since patient comfort represents a major determinant for the success of a non-invasive respiratory support, especially when patient tolerance and compliance are challenged by the extended length of the treatment, we set up the present pilot study aiming at assessing patient comfort during oxygen support with asymmetrical HFNCs, comparing two cannula sizes, one completely occluding the nostril and one a size smaller.

Secondary outcome variables include patient dyspnea, lung aeration, as assessed with electrical impedance tomography (EIT), ventilatory efficiency, and gas exchange.

Measurements During HFNC support, the FiO2 will be titrated to maintain a peripheral oxygen saturation between 90% and 94%, the gas flow rate will be set at 50-60 L/min, and the temperature of the heated humidifier (Fisher&Paykel Healthcare, New Zealand) will be set at 37° C (absolute humidity delivered 44 mgH2O/L) for the entire study period.

The following parameters will be measured during the last 10 minutes of each step:

Comfort, assessed by a 0-10 numeric rating scale (NRS); Dyspnea, assessed by the Borg scale; Lung aeration, assessed by EIT. In detail, a 16-electrode EIT belt will be placed around the chest, as previously described. The following EIT parameters will be recorded: (i) the average global tidal volume (VT) and the percentage of VT distributed to non-dependent and dependent lung regions (VTglob, VTnon-dep, and VTdep, respectively); (ii) the minute ventilation (MV) and the corrected MV, calculated as [(VTglob x PaCO2)/40 mmHg]* respiratory rate per minute- 1, where 40 mmHg is the ideal value of PaCO2; (iii) the global and regional changes in end-expiratory lung impedance (EELI) (estimating end-expiratory lung volume) (ΔEELIglob, ΔEELInon-dep, and ΔEELIdep, respectively); (iv) the global inhomogeneity index (GI) and the regional ventilation delay (RVD); Respiratory rate, SpO2, pH, arterial partial pressure of carbon dioxide (PaCO2), arterial partial pressure of oxygen (PaO2), arterial partial pressure of oxygen to fraction of inspired oxygen ratio (PaO2/FiO2), and ventilatory ratio.

ELIGIBILITY:
Inclusion Criteria:

- adult patients (>18 years old) requiring oxygen support in the ICU

Exclusion Criteria:

* pregnancy;
* presence of tracheostomy;
* contraindications to EIT;
* contraindications to HFNCs positioning,
* clinical evidence of nare occlusion (patient will be asked to deeply inspire from the nose while researcher occludes manually each nostril alternately: if unable to breath from the free nare with the other one occluded, patient will not be eligible for participating to the study), or very small nare fitting only the S-sized Duet cannulas;
* patients requiring nasogastric tubes for mandatory clinical reasons, i.e., delayed gastric emptying, upper abdominal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to the ICU and requiring oxygen support for any reason.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
COMFORT | After 60 minutes of HFNC support
  The present pilot study aims at assessing patient comfort during oxygen support with asymmetrical HFNCs, comparing two cannula sizes, one completely occluding the nostril and one a size smaller. The evaluation scale is the 0-10 numeric rating scale (NRS).
  Each step will be 60 min long and a 10-min 'wash-out' phase with Venturi mask support will be required before each step.

SECONDARY OUTCOMES:
DYSPNEA | After 60 minutes of HFNC support
  The present pilot study aims at assessing patient dyspnea, measured by the BORG scale [8] during oxygen support with asymmetrical HFNCs, comparing two cannula sizes, one completely occluding the nostril and one a size smaller.
  Each step will be 60 min long and a 10-min 'wash-out' phase with Venturi mask support will be required before each step.
LUNG AERATION | After 60 minutes of HFNC support
  The present pilot study aims at assessing LUNG AERATION, measured by electrical impedance tomography (EIT), during oxygen support with asymmetrical HFNCs, comparing two cannula sizes, one completely occluding the nostril and one a size smaller.
  Each step will be 60 min long and a 10-min 'wash-out' phase with Venturi mask support will be required before each step.
Respiratory rate, peripheral oxygen saturation, gas-changes, ratio between PaO2 and inspiratory oxygen fraction, ventilatory ratio [10] | After 60 minutes of HFNC support
  The present pilot study aims at assessing respiratory rate, peripheral oxygen saturation, gas-changes, ratio between PaO2 and inspiratory oxygen fraction and ventilatory ratio, during oxygen support with asymmetrical HFNCs, comparing two cannula sizes, one completely occluding the nostril and one a size smaller.
  Each step will be 60 min long and a 10-min 'wash-out' phase with Venturi mask support will be required before each step.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto di Anestesia e Rianimazione, ISTAR 3, Padua, Italy
  - Azienda Ospedale Università Padova, Padua, Padova

IPD SHARING:
Plan to Share IPD: No